CLINICAL TRIAL: NCT06354439
Title: Use of Letrozole in the Treatment of Early Ectopic Pregnancy
Brief Title: Use of Letrozole for Ectopic Pregnancy
Acronym: EcZOL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 77015224.6.1001.5327
Record Dates: First submitted 2024-04-01; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Ectopic Pregnancy
Keywords: ectopic pregnancy; letrozole; methotrexate
MeSH Terms: conditions — Pregnancy, Ectopic | interventions — Letrozole; Methotrexate

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Masking Description: Due to the nature of the outcome and the interventions, blinding was not considered an issue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- letrozole (Experimental): Patients will receive 10mg of letrozole por 7 days.
  Interventions: Drug: Letrozole tablets
- Methotrexate (Active Comparator): Patients will receive a single intramuscular dose of 100 mg of methotrexate.
  Interventions: Drug: Methotrexate Sodium

INTERVENTIONS:
Drug: Letrozole tablets — 10 mg of letrozole PO for 7 days
  Other Names: letrozole 2,5mg - 4 tables
  Arms: letrozole
Drug: Methotrexate Sodium — 100 mg of methotrexate IM, single dose
  Other Names: methotrexate intramuscular (IM)
  Arms: Methotrexate

SUMMARY:
A randomized clinical trial using oral letrozole 10mg/day for 7 days, for treating early cases of ectopic pregnancy, compared to intramuscular methotrexate

DETAILED DESCRIPTION:
This is a multicenter randomized clinical trial on the use of letrozole in the medical treatment of tubal ectopic pregnancy. Tubal ectopic pregnancy is an abnormal pregnancy in the fallopian tube. They occurred in about 8% of all pregnancies presenting to the emergency department. Methotrexate (MTX), administered systemically (intramuscularly), is a widely used medication for the treatment of unruptured tubal ectopic pregnancies and has been recommended as first-line treatment for early cases of ectopic pregnancy.

Letrozole is an aromatase inhibitor and can suppress estradiol levels. Some recent studies have shown that its use can be applied in cases of ectopic pregnancy.

The aim of this non-inferiority clinical trial is to verify that letrozole treatment is non-inferior to methotrexate treatment in women with early ectopic pregnancy who are hemodynamically stable.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Diagnosis of ectopic pregnancy
* Desire for reproduction
* Ease of return
* Undetermined pregnancy location with abnormal hCG growth
* Presence of a heterogeneous adnexal mass on pelvic ultrasound suggestive of a tubal ectopic pregnancy with an hCG level ≤ 3000 mIU/ml
* Absence of fetal cardiac activity
* Average diameter of the adnexal mass ≤ 3.5 cm
* Hemodynamically stable
* No significant abdominal pain (i.e, < 6 on a visual analog scale)

Exclusion Criteria:

* Presence of a significant amount of free fluid in the pelvis (as assessed by the ultrasound technician)
* Allergy to methotrexate or letrozole
* A reduction in β-hCG ≥ 50% in 2 measurements with 48 hours between them or

  ≥ 85% in 4 days, or ≥ 95% in 7 days before randomization
* Abnormal liver function test (Alanine transaminase (ALT) ≥ 2 times the upper limit of normal)
* Abnormal renal function test (glomerular filtration rate ≤ 45 ml/min)
* Hemoglobin <10 g/dl
* Platelets <120.000/ml
* Presence of heterotopic pregnancy
* Do not wish to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — ciswomen with ectopic pregnancy.
Enrollment: 130 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
levels of beta fraction of human chorionic gonadotropin (beta-hCG) | weekly after the first day of intervention until reaching levels of beta-hCG below 5 milli-International unit per milliliter (assessed up to 5 months)"
  On day 4 (D4) and 7(D7), beta-hCG levels will be measured. If a reduction equal or above 15% between D4 and D7 were observed, serum beta-hCG will be measured until reach levels < 5 milli-International unit per milliliter (mIU/ml).

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo F Savaris, MD, PhD, Study Chair — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All collected anonymized data will available so others may reproduce the results
Supporting Information: Study Protocol
Time Frame: march 28, 2024 until march 28 2044
Access Criteria: open access
URL: https://docs.google.com/document/d/14oXyHS7InjCzTCvQW78Lf6pjgLmRb5HBB8otBDl87x0/edit?usp=sharing

REFERENCES:
- [Background] Link CA, Maissiat J, Mol BW, Barnhart KT, Savaris RF. Diagnosing ectopic pregnancy using Bayes theorem: a retrospective cohort study. Fertil Steril. 2023 Jan;119(1):78-86. doi: 10.1016/j.fertnstert.2022.09.016. Epub 2022 Oct 26. PMID 36307292
- [Background] Farquhar CM. Ectopic pregnancy. Lancet. 2005 Aug 13-19;366(9485):583-91. doi: 10.1016/S0140-6736(05)67103-6. PMID 16099295
- [Background] Bouyer J, Coste J, Fernandez H, Pouly JL, Job-Spira N. Sites of ectopic pregnancy: a 10 year population-based study of 1800 cases. Hum Reprod. 2002 Dec;17(12):3224-30. doi: 10.1093/humrep/17.12.3224. PMID 12456628
- [Background] van Mello NM, Mol F, Ankum WM, Mol BW, van der Veen F, Hajenius PJ. Ectopic pregnancy: how the diagnostic and therapeutic management has changed. Fertil Steril. 2012 Nov;98(5):1066-73. doi: 10.1016/j.fertnstert.2012.09.040. PMID 23084008
- [Background] Diagnosis and Management of Ectopic Pregnancy: Green-top Guideline No. 21. BJOG. 2016 Dec;123(13):e15-e55. doi: 10.1111/1471-0528.14189. Epub 2016 Nov 3. No abstract available. PMID 27813249
- [Background] Qian X, Li Z, Ruan G, Tu C, Ding W. Efficacy and toxicity of extended aromatase inhibitors after adjuvant aromatase inhibitors-containing therapy for hormone-receptor-positive breast cancer: a literature-based meta-analysis of randomized trials. Breast Cancer Res Treat. 2020 Jan;179(2):275-285. doi: 10.1007/s10549-019-05464-w. Epub 2019 Oct 12. PMID 31606823
- [Background] Casper RF, Mitwally MF. Use of the aromatase inhibitor letrozole for ovulation induction in women with polycystic ovarian syndrome. Clin Obstet Gynecol. 2011 Dec;54(4):685-95. doi: 10.1097/GRF.0b013e3182353d0f. PMID 22031258
- [Background] Auger N, Ayoub A, Wei SQ. Letrozole: future alternative to methotrexate for treatment of ectopic pregnancy? Fertil Steril. 2020 Aug;114(2):273-274. doi: 10.1016/j.fertnstert.2020.04.063. Epub 2020 Jul 1. No abstract available. PMID 32622661
- [Background] Mitwally MF, Hozayen WG, Hassanin KMA, Abdalla KA, Abdalla NK. Aromatase inhibitor letrozole: a novel treatment for ectopic pregnancy. Fertil Steril. 2020 Aug;114(2):361-366. doi: 10.1016/j.fertnstert.2020.04.001. Epub 2020 Jul 1. PMID 32622660
- [Background] Rezaei Z, Ghaemi M, Feizabad E, Ghavami B, Akbari Asbagh F, Davari Tanha F, Ebrahimi M, Khalaj Sereshki Z. The Effective Role of Adding Letrozole to Methotrexate in the Management of Tubal Ectopic Pregnancies, a Randomized Clinical Trial. Iran J Pharm Res. 2021 Fall;20(4):378-384. doi: 10.22037/ijpr.2021.115659.15461. PMID 35194453
- [Background] Alabiad MA, Said WMM, Gad AH, Sharaf ElDin MTA, Khairy DA, Gobran MA, Shalaby AM, Samy W, Abdelsameea AA, Heraiz AI. Evaluation of Different Doses of the Aromatase Inhibitor Letrozole for the Treatment of Ectopic Pregnancy and Its Effect on Villous Trophoblastic Tissue. Reprod Sci. 2022 Oct;29(10):2983-2994. doi: 10.1007/s43032-022-00993-0. Epub 2022 Jun 14. PMID 35701686
- [Background] Lipscomb GH, Gomez IG, Givens VM, Meyer NL, Bran DF. Yolk sac on transvaginal ultrasound as a prognostic indicator in the treatment of ectopic pregnancy with single-dose methotrexate. Am J Obstet Gynecol. 2009 Mar;200(3):338.e1-4. doi: 10.1016/j.ajog.2008.12.006. PMID 19254596